CLINICAL TRIAL: NCT00366613
Title: Clinical Evaluation of the Use of Sealed Capsule Irrigation With Sodium Chloride During Pediatric Cataract Surgery and IOL Implantation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: We wish to wait until there is more data available using this substance.
Sponsor: Medical University of South Carolina (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SEI-06-002
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2007-08

CONDITIONS: Cataract Extraction
Keywords: Cataract; Cataract Extraction
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction; Sodium Chloride

INTERVENTIONS:
Procedure: Cataract surgery with Perfect Capsule and Sodium Chloride

SUMMARY:
This study involves using both a device that seals the capsular bag (where the lens is located) allowing safer irrigation of the capsular bag and sodium chloride to irrigate the capsular bag during cataract surgery on children. The purpose of this study is to determine if the use of the device, Perfect Capsule, along with sodium chloride reduces the development of posterior capsule opacification (PCO), a possible complication of cataract surgery. PCO is the clouding of the rear portion of the natural membrane or capsule that holds the artificial lens. It requires additional procedures to correct the problem. Sodium chloride is not usually used during cataract surgery. It will be used to irrigate the capsular bag and remove any residual cells that contribute to the development of PCO. Perfect Capsule will prevent the sodium chloride from touching other parts of the eye. The goal of this study is to determine if irrigation with sodium chloride will lower the incidence of PCO after cataract surgery.

DETAILED DESCRIPTION:
Dramatic advances have occurred in the treatment of childhood cataracts in the last 10 years. Intraocular lens implantation (IOL) has been universally accepted as standard of care in children beyond 2 years of age. Despite advances in cataract surgery in children, PCO remained a significant complication following pediatric cataract surgery. In addition to being visually disturbing, it also induces amblyopia in children and if not treated at earliest, irreversible visual changes may occur. The younger the child, more acute is the problem: PCO occurs faster and effect of amblyopia is more pronounced. PCO generally requires second surgical intervention, as closure of the opening made by YAG capsulotomy is very common after pediatric cataract surgery. Many times, children are not cooperative to sit down for YAG capsulotomy, and that may also be an additional indication for second surgery for PCO.

Removal of residual epithelial cells is one of the key factors to avoid the complication of PCO. Several chemicals have been suggested in experimental settings to remove or kill these residual lens epithelial cells. However, they are toxic to other ocular structures. Researchers are searching for a device which can help to selectively kill these lens epithelial cells. In the long term, this may help to avoid PCO.

Perfect Capsule: Perfect CapsuleTM (Milvella ltd) is a sterile single use ophthalmic instrument used to perform sealed irrigation of the capsular bag during cataract surgery in order to facilitate irrigation of the capsule without the irrigation fluid contacting other ocular structures. The device has the FDA approval via 510(k) in the USA, and is CE marked in Europe. No specific age limit has been listed for FDA approval. The device (see fig) consists of a 7 mm diameter head, a 3 mm wide body and a 4 mm wide foot that remains external to the eye. The head of the device comprises a circumferential vacuum channel connected to a vacuum syringe via a vacuum tube. The central portion of the head forms a plug with an irrigation/aspiration (I/A) channel (the body) which extend through the cornea allowing fluids to be injected into the under surface of the plug and thus into the capsule. The device has an internal diameter of 5 mm, is molded in medical grade silicone, packaged and gamma sterilized. It can be easily rolled or folded to pass through the standard corneal incision into the eye and positioned on the anterior surface of the capsule using standard ophthalmic instrument.

Concentrated Sodium Chloride: Concentrated Sodium Chloride injection, USP 23.4% (American Regent Laboratories, Inc., Shirley, NY) is sterile, preservative free, nonpyrogenic solution of Sodium Chloride in water for injection. Deionised water has been shown to lyse lens epithelial cells through osmotic flow. Concentrated Sodium Chloride is not currently indicated for intraocular use and is also expected to affect the corneal endothelium. Use of Perfect Capsule will help to avoid the contact of Concentrated sodium Chloride to the endothelial cells.

For the purpose of this study, Concentrated Sodium Chloride for injection will be colored with minimal fluorescein so that the flow and location of it can be visualized throughout the procedure. Viscoelastic within the anterior chamber will provide additional protection for the corneal endothelium.

SCI with Perfect Capsule and Concentrated Sodium Chloride: Perfect CapsuleTM allows for the empty capsular bag to be irrigated with Concentrated Sodium Chloride. A previous study in rabbits has shown that toxic solutions can be safely used for SCI. It has also been shown that the irrigation solution is contained within the capsular bag when SCI is performed in humans. Dr. Auffarth has presented a summary of the two year Australian study results and one year European multi-center clinical trial results performing SCI with distilled water in humans (At American Society of Cataract and Refractive Surgery meeting, 2005). In 44 patients studied, the system could be used without complication and the endothelial cell count and corneal pachymetry was not different from the control eyes. Visual acuity development over a 6-12 months period was similar in both groups. Retro-illumination photographs showed a higher incidence of fibrosis and anterior capsule whitening in the control group compared to the SCI group. With the currently available IOLs, PCO is not a significant complication in adult eyes at 1-2 year postoperative period. Long-term results will be needed to detect the difference (if any) in terms of PCO in adult eyes. In contrast, PCO is a significant problem in pediatric eyes. It occurs at a much faster rate and during early postoperative period in children's eyes as compared to adult's eyes. Younger the child at the time of cataract surgery, more acute is the problem. Thus, it is possible to see the difference in terms of PCO (if any) with the use of Perfect Capsule in children's eyes during early postoperative period, as 1 year postoperatively in this study. We are not aware of any published results or results presented at the meeting showing use of SCI or distilled water in pediatric eyes.

ELIGIBILITY:
Inclusion Criteria:

* bilateral cataract
* 4 - 18 years of age
* Informed consent from the parents/legal guardian.

Exclusion Criteria:

* traumatic cataract
* fellow eye - visually not significant cataract
* fellow eye surgery not planned during the study enrollment period
* weak or compromised posterior or anterior capsule
* dense posterior capsule plaque
* preexisting posterior capsule defect
* capsulorhexis diameter>5 mm
* radial capsular tears
* defects within the remaining capsular bag
* inability to visualize the entire capsulorhexis
* shallow anterior chamber
* very high vitreous pressure

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2005-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marion E Wilson, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Storm Eye Institute, Medical University of South Carolina, Charleston, South Carolina, United States